CLINICAL TRIAL: NCT02833272
Title: Deprescribing Sedative Hypnotics on the Clinical Teaching Unit Using a Patient Empowerment Tool
Brief Title: Understanding Benzodiazepine and Non-benzodiazepine Sedative Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Todd Lee, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-372
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Frailty; Deprescription; Aged
Keywords: benzodiazepines; Z-drugs
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EMPOWER Educational Brochure (Experimental): This is the only arm of the study. All participants will undergo the intervention, which is an educational brochure (EMPOWER educational brochure) to explain the possible harms of benzodiazepine and non-benzodiazepine sedative drugs.
  Interventions: Behavioral: EMPOWER Educational Brochure

INTERVENTIONS:
Behavioral: EMPOWER Educational Brochure — The EMPOWER educational brochure explains the risk of benzodiazepine and non-benzodiazepine sedative use to patients with a current prescription. The brochure also provides a tapering schedule if the patient chooses to discontinue taking the drug.

SUMMARY:
Inappropriate medication use among the elderly ranges from 11% to 62% and is a major concern for patient safety. Benzodiazepines account for approximately 20 to 25% of inappropriate medications prescribed to the elderly, thus reducing their inappropriate use could have a substantial impact on patient safety and overall well-being among elderly patients. The Choosing Wisely Canada- Geriatrics guidelines for high value health care recommend against the prescription of benzodiazepines or other sedative-hypnotics (Z drugs) in older adults as first choice for insomnia, agitation or delirium. Despite evidence of potential harms, benzodiazepines and non-benzodiazepine sedatives (including the "Z-drugs": eszopiclone, zopiclone, zolpidem and zaleplon, henceforth referred to as "sedatives") continue to be prescribed inappropriately to patients in hospital and community settings.

Our primary objective is to facilitate the deprescription of benzodiazepine and non-benzodiazepine sedative hypnotics (sedatives) using a combination of physician education sessions and an updated patient educational pamphlet based on Tannenbaum's EMPOWER study conducted in a community-based setting.

DETAILED DESCRIPTION:
This study will be a pragmatic before-after intervention trial at the McGill University Health Centre (MUHC) Royal Victoria Hospital (Glen Site) using historical controls from 2014-2016 at our hospital.The intervention will begin July 2016 and conclude January 2016.

The intervention will include the following components:

1. Educational campaign toward physicians about benzodiazepine and Z-drug prescriptions:

   An educational campaign about the purpose of the study and risks of benzodiazepine and sedative prescriptions will be delivered to physicians in each intervention cluster. The educational campaign will include a presentation by the chief of the medical service at teaching rounds at the beginning of the intervention, an electronic message sent to all physicians on the medical service, and posting of the Choosing Wisely Canada- Geriatrics guidelines.
2. In-hospital patient education campaign:

Patients will be identified from the pharmacy database and validated by a research associate in collaboration with the unit pharmacists based on the patient's best possible medication history taken at time of admission. Eligibility will be confirmed by the patient's treating physician with support from the principal investigator and site coordinators. Patients will receive a previously validated (in the outpatient setting) educational brochure about the risks of chronic sedative use and how to stop using them through a tapering regimen. The booklet currently includes information about benzodiazepines but will be adapted to also include information about sedatives. The preparation of the brochure has been validated in both English and French for comprehension and readability.

Clusters will be defined by clinical teaching unit (CTU) at the Royal Victoria Hospital, - the C9 CTU and D9 CTU. Follow up of discharged patients will be until 30 and 90 days post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients 65 years or older admitted to study units
* Have a benzodiazepine or sedative prescription used at least 3 times in the week prior to enrolment

Exclusion Criteria:

* Less than 65 years of age
* Admitted for the treatment of alcohol or benzodiazepine withdrawal
* Not having a prescription for benzodiazepines or Z-drugs
* Not reporting use of either medication at least 3 times in the week prior to admission
* Not being enrolled in the provincial drug plan
* Opting out of the provincial drug database (DSQ)
* Previous enrolment in the study
* Patients expected to die before primary endpoint can be realized (e.g., patients admitted for end of life care or prognosis of 3 months or less)
* Patient lives in nursing home and has dementia without an identifiable proxy
* Inability for patient or proxy to speak English or French
* No means of contacting patient or proxy after discharge

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Stopped Use | 90 days post-discharge
  Investigators will evaluate whether the patient has stopped use of benzodiazepines within 90 days of discharge from the hospital.

SECONDARY OUTCOMES:
Sleep disturbance: sleep quality assessed by the PROMIS Sleep Disturbance 4a Short Form | 90 days post-discharge
  Investigators will evaluate whether the patient's sleep quality has changed since they left the hospital. The PROMIS Sleep Disturbance 4a Short Form will be used to assess sleep.
Change in patient self-reported falls | 90 days post-discharge
  Investigators will evaluate whether there has been any change in patient self-reported falls.

CONTACTS AND LOCATIONS:
Overall Officials: Emily G McDonald, MD MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre (Royal Victoria Hospital), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Tannenbaum C, Martin P, Tamblyn R, Benedetti A, Ahmed S. Reduction of inappropriate benzodiazepine prescriptions among older adults through direct patient education: the EMPOWER cluster randomized trial. JAMA Intern Med. 2014 Jun;174(6):890-8. doi: 10.1001/jamainternmed.2014.949. PMID 24733354
- [Background] Guaraldo L, Cano FG, Damasceno GS, Rozenfeld S. Inappropriate medication use among the elderly: a systematic review of administrative databases. BMC Geriatr. 2011 Nov 30;11:79. doi: 10.1186/1471-2318-11-79. PMID 22129458
- [Background] Brekke M, Rognstad S, Straand J, Furu K, Gjelstad S, Bjorner T, Dalen I. Pharmacologically inappropriate prescriptions for elderly patients in general practice: How common? Baseline data from The Prescription Peer Academic Detailing (Rx-PAD) study. Scand J Prim Health Care. 2008;26(2):80-5. doi: 10.1080/02813430802002875. PMID 18570005
- [Background] van der Hooft CS, Jong GW, Dieleman JP, Verhamme KM, van der Cammen TJ, Stricker BH, Sturkenboom MC. Inappropriate drug prescribing in older adults: the updated 2002 Beers criteria--a population-based cohort study. Br J Clin Pharmacol. 2005 Aug;60(2):137-44. doi: 10.1111/j.1365-2125.2005.02391.x. PMID 16042666
- [Background] American Geriatrics Society 2012 Beers Criteria Update Expert Panel. American Geriatrics Society updated Beers Criteria for potentially inappropriate medication use in older adults. J Am Geriatr Soc. 2012 Apr;60(4):616-31. doi: 10.1111/j.1532-5415.2012.03923.x. Epub 2012 Feb 29. PMID 22376048
- See also: Choosing Wisely Canada - Canadian Geriatrics Society Recommendations — http://www.choosingwiselycanada.org/recommendations/geriatrics/